

| BI Study Number: | 1403-0024 |
|---|---|
| Title: Demographic, clinical characteristics, and treatment outco associated with dedifferentiated liposarcoma patients in Cartesian Ca | |
| NCT number: | NCT06115681 |
| Date: | October 9, 2023 |

This page has been added to the Statistical and Epidemiological Analysis Plan (SEAP) to reflect the requirements by ClinicalTrials.gov. This information is not part of the standard document.



# STATISTICAL AND EPIDEMIOLOGICAL ANALYSIS PLAN (SEAP)

| <b>Document Number:</b> | c43137559 |
|---|---|
| BI Study Number: | 1403-0024 |
| BI Investigational<br>Product | Not applicable |
| Title: | Demographic, clinical characteristics, and treatment outcomes associated with dedifferentiated liposarcoma patients in China |
| Brief lay title: | Real-world study of dedifferentiated liposarcoma patients in China |
| SEAP version identifier: | 1.0 |
| Date of last version of SEAP: | NA |
| ONIS Statistician | |
| [SEAP author] | |
| ONIS | |
| [SEAP reviewer] | |
| ONIS Data | |
| [SEAP reviewer] | |

Proprietary confidential information

© 2023 Boehringer Ingelheim Group of companies. All rights reserved.

This document may not - in full or in part - be passed on, reproduced, published or otherwise used without prior written permission

Statistical and Epidemiological Analysis Plan (SEAP) for Observational and Non-Interventional Studies (ONIS)


### **TABLE OF CONTENTS**

| 1. LIST OF ABBREVIATIONS | 3 |
|-----------------------------------------|-----|
| 2. RESPONSIBLE PARTIES | 3 |
| 3. PURPOSE AND SCOPE | |
| 4. AMENDMENTS AND UPDATES | 4 |
| 5. RESEARCH QUESTION AND OBJECTIVES | . 4 |
| 6. RESEARCH METHODS | 4 |
| 6.1 STUDY DESIGN | 4 |
| 6.2 SETTING | 5 |
| 6.3 STUDY POPULATION | 5 |
| 6.4 STUDY VISITS | |
| 7. VARIABLES | . 6 |
| 7.1 OUTCOMES | . 7 |
| 7.1.1 Primary outcomes | 7 |
| 7.1.2 Secondary outcomes | 7 |
| 8. DATA SOURCES | |
| 9. DATA MANAGEMENT AND SOFTWARE/TOOLS | 15 |
| 9.1 SOURCE DATA | 15 |
| 9.2 DATA CURATION | |
| 9.3 SOFTWARE/TOOLS | |
| 9.4 HANDLING OF MISSING VALUES | |
| 10. DATA ANALYSIS | 16 |
| 10.1 MAIN ANALYSIS | 17 |
| 10.1.1 Analysis of primary objective | |
| 10.1.2 Analysis of secondary objectives | 17 |
| 10.3 SAFETY ANALYSIS | |
| 11. QUALITY CONTROL | 19 |
| 12. REFERENCES | 19 |
| 12.1 PUBLISHED REFERENCES | 19 |
| 12.2 UNPUBLISHED REFERENCES | 19 |
| ANNEX 1. ADDITIONAL INFORMATION | 20 |
| ANNEY 2 MOCK TADI E AND FIGURE | 20 |

Statistical and Epidemiological Analysis Plan (SEAP) for Observational and Non-Interventional Studies (ONIS) 

### 1. LIST OF ABBREVIATIONS

| 1L | First line |
|----|-------------|
| 2L | Second line |
| 3L | Third line |

BI Boehringer Ingelheim

CDC Center for Disease Control and Prevention Center

CI Confidence Interval CRF Case report form

CSCO Chinese Society of Clinical Oncology

DDLPS Dedifferentiated liposarcoma

ECOG Eastern Cooperative Oncology Group

EMPI Enterprise Master Patient Index

EMR Electronic medical records

GPP Good Pharmacoepidemiology Practice

HCRU Healthcare resource utilization IEC Independent Ethics Committee

IQR Interquartile range KM Kaplan-Meier LOT Line of therapy

NATDSS National Anti-Tumor Drug Surveillance System

NCC National Cancer Center

NCCN National Comprehensive Cancer Network

NIS Non-Interventional Study

ONIS Observational and Non-Interventional Study

OS Overall survival

SAS Statistical Analysis System

SD Standard deviation

SEAP Statistical and Epidemiological Analysis Plan

SOP Standard operating procedure

### 2. RESPONSIBLE PARTIES

Observational and Non-Interventional Study (ONIS) Statistician:

•

#### SEAP reviewers are:

- Boehringer Ingelheim (BI) ONIS
- ONIS Line
- Global TM Epi:

Statistical and Epidemiological Analysis Plan (SEAP) for Observational and Non-Interventional Studies (ONIS)


| • | Global Medical Advisor: |
|---|-------------------------|
| • | PSTAT: |
| • | ABRT |
| • | Global TA Epi: |
| • | ONIS Data |

#### 3. PURPOSE AND SCOPE

This ONIS is conducted based on existing database. This document provides an overview of the processes and procedures of data quality review and management, methods used to describe, analyze and display data, and quality control of data throughout the conduct of ONIS.

### 4. AMENDMENTS AND UPDATES

Not applicable.

### 5. RESEARCH QUESTION AND OBJECTIVES

### **Primary objective:**

To describe the overall survival (OS) of Chinese unresectable locally advanced or metastatic dedifferentiated liposarcoma (DDLPS) patients

### **Secondary objective:**

To describe the treatment patterns of Chinese DDLPS patients

### **Exploratory objective:**

To describe demographic, clinical characteristics and treatment outcomes of Chinese DDLPS patients

To describe the direct medical cost and healthcare resource utilization of Chinese DDLPS patients

### 6. RESEARCH METHODS

#### 6.1 STUDY DESIGN

This will be a non-interventional/observational study of Chinese DDLPS patients using existing data curated by . No BI product will be studied, and no new interventions or procedures will be performed.

The primary outcome is OS. Secondary outcomes include survival after initial diagnosis, and treatment patterns. Exploratory outcomes may include patient demographics, clinical characteristics, duration of treatment (DOT), time to next treatment (TTNT) by lines,

Statistical and Epidemiological Analysis Plan (SEAP) for Observational and Non-Interventional Studies (ONIS)


healthcare resource utilization and direct medical cost, etc. None of the outcomes reflect safety issues.

#### 6.2 SETTING

In this study, patient data from NATDSS network from January 1, 2013 to December 31, 2022 will be used. Details of data source are described in section 8.

#### **6.3 STUDY POPULATION**

Inclusion criteria:

- Patient has two or more documented clinical visits in the National Anti-Tumor Drug Surveillance System (NATDSS) network on or after January 1, 2013.
- Patient has a confirmed diagnosis of DDLPS during his/her lifetime.
- At least 18 years old at the date of initial diagnosis

No exclusion criteria are applied.

Eligible population will be divided into two groups:

- Cohort 1 will include unresectable locally advanced or metastatic DDLPS patients who received at least one line of systemic antineoplastic treatment by the end of cohort identification period (index date = start date of first line (1L) treatment).
- Cohort 2 will include patients with DDLPS who have not initiated 1L systemic antineoplastic treatment by the end of cohort identification period (index date = date of initial DDLPS diagnosis during cohort identification period). Patients initiated 1L treatment afterwards or patients received adjuvant and/or neoadjuvant therapy only through follow-up will be included in Cohort 2.

In both cohorts, 1L therapy will be defined as the initial set of drugs used after unresectable locally advanced or metastatic diagnosis. Metastatic patients will be defined as those with metastatic diagnosis or presence of metastatic sites; unresectable locally advanced patients will be defined as those with advanced diagnosis and without subsequent surgical resection.

### 6.4 STUDY VISITS

Definitions of relevant time periods are detailed below.

Study period: January 1, 2013 – December 31, 2022

Baseline period: All available data prior to index date

**Cohort identification period:** January 1, 2013 – December 31, 2021 (one year before end of study period)

Statistical and Epidemiological Analysis Plan (SEAP) for Observational and Non-Interventional Studies (ONIS)

**Index date:** The index date for Cohort 1 will set to the date of initiation of 1L treatment; the index date for Cohort 2 will be the date of initial DDLPS diagnosis during cohort identification period.

**Follow-up period:** From index date until date of death, if available, or the date of censoring if there is no record of death, whichever occurs first. For survival and treatment patterns, the date of censoring will be the last activity date, defined as the date of the last visit of any type prior to the end of the study period.

Figure 1 illustrates the time periods for the study timelines.

#### (a). Cohort 1



#### (b). Cohort 2



Figure 1. Overall study period

Abbreviations: 1L = first line

### 7. VARIABLES

The analysis will be descriptive only, and there are no *a priori* hypotheses. There will be no prespecified exposures or covariates to be used as the basis for formal statistical testing and for *a priori* comparison of groups.

Statistical and Epidemiological Analysis Plan (SEAP) for Observational and Non-Interventional Studies (ONIS)


#### 7.1 OUTCOMES

### 7.1.1 Primary outcomes

### OS

Outcome type: PrimaryOutcome name: OS

• Time frame: Time from index date until the earliest record of death or end of the study

period

■ **Population:** Cohort 1

OS as an event for each patient in Cohort 1 will be defined as the date of death minus the index date or the start day of each line of therapy (LOT). For patients with no record of death, OS will be censored at the last activity date before the end of the study period.

### 7.1.2 Secondary outcomes

### Survival after initial diagnosis

Outcome type: Secondary

• Outcome name: Survival after initial diagnosis

• **Time frame**: Time from initial diagnosis until the earliest record of death or end of the study period

• **Population**: Cohort 1, Cohort 2

Survival after initial diagnosis for each patient will be defined as the date of death minus the date of initial diagnosis. For patients with no record of death, survival after initial diagnosis will be censored at the last activity date before the end of the study period.

### Description of treatment patterns

Outcome type: Secondary

• Outcome name: Treatment patterns

• Time frame: Treatment patterns are assessed at the index date and during follow-up

■ **Population**: Cohort 1, Cohort 2

The following variables of interest will be assessed to describe treatment patterns defined by LOT and regimens.

Treatment patterns by LOT and regimens

| Variable | Definition | Timing |
|---|---|---|
| 1L Treatment Type | Regimen name from LOT data for treatments with line number = 1, 2 and 3. Treatment | Any time after |
| 2L Treatment Type | types will be classified as follows, specific treatments and categories may change upon examination of the data: | index date |
| 3L Treatment Type | | |

Statistical and Epidemiological Analysis Plan (SEAP) for Observational and Non-Interventional Studies (ONIS)

| Variable | Definition | Timing |
|---|---|---|
| | NCCN/CSCO preferred | |
| | <ul> <li>Doxorubicin</li> </ul> | |
| | <ul> <li>Epirubicin</li> </ul> | |
| | <ul> <li>Liposomal doxorubicin</li> </ul> | |
| | AD (doxorubicin, dacarbazine) | |
| | <ul> <li>AIM (doxorubicin, ifosfamide, mesna)</li> </ul> | |
| | Ifosfamide, epirubicin, mesna | |
| | <ul> <li>Larotrectinib (NTRK fusion pos sarcomas only)</li> </ul> | |
| | <ul> <li>Entrectinib (NTRK fusion pos sarcomas only)</li> </ul> | |
| | <ul> <li>Pazopanib</li> </ul> | |
| | • Eribulin | |
| | Trabectedin | |
| | Other | |
| | <ul> <li>AD LMS only (doxorubicin,<br/>dacarbazine)</li> </ul> | |
| | Gemcitabine and docetaxel | |
| | Gemcitabine | |
| | Gemcitabine and vinorelbine | |
| | Gemcitabine and dacarbazine | |
| | <ul> <li>Dacarbazine</li> </ul> | |
| | <ul> <li>Ifosfamide</li> </ul> | |
| | Temozolomide | |
| | Vinorelbine | |
| | <ul> <li>Regorafenib</li> </ul> | |
| | <ul> <li>MAID (mesna, doxorubicin, ifosfamide, dacarbazine)</li> </ul> | |
| | <ul> <li>Pembrolizumab</li> </ul> | |
| | <ul> <li>durvalumab</li> </ul> | |
| | • Other | |
| Total number of treatment lines | From LOT data, for all lines after index date, categorical variable defined as total of treatment lines reported. | Any time after index date |
| Concurrent steroid therapy | Any record of a drug classified as a corticosteroid. | Anytime from the start to end of 1L, 2L, or 3L |

Statistical and Epidemiological Analysis Plan (SEAP) for Observational and Non-Interventional Studies (ONIS)


| Variable | Definition | Timing |
|---|---|---|
| Concurrent | Any record of a drug classified as an | Anytime from the |
| immunosuppressant | immunosuppressant therapy. | start to end of 1L, |
| therapy | | 2L, or 3L |
| Concurrent | Any record of a drug classified as a hormone | Anytime from the |
| hormone | replacement therapy. | start to end of 1L, |
| replacement therapy | | 2L, or 3L |

Abbreviations: 1L = first line; 2L = second line; 3L = third line; CSCO = Chinese Society of Clinical Oncology; LOT = line of therapy; NCCN = National Comprehensive Cancer Network



Property of Boehringer Ingelheim Group of Companies - Use current version only and according to confidentiality principles

Statistical and Epidemiological Analysis Plan (SEAP) for Observational and Non-Interventional Studies (ONIS)




Statistical and Epidemiological Analysis Plan (SEAP) for Observational and Non-Interventional Studies (ONIS)




Statistical and Epidemiological Analysis Plan (SEAP) for Observational and Non-Interventional Studies (ONIS)




Statistical and Epidemiological Analysis Plan (SEAP) for Observational and Non-Interventional Studies (ONIS)




Statistical and Epidemiological Analysis Plan (SEAP) for Observational and Non-Interventional Studies (ONIS)




### 8. DATA SOURCES

will develop a custom, curated dataset for this study based on longitudinal electronic medical records (EMR) data from the NATDSS, the largest cancer registry database in China. This database, established in 2018 by China National Cancer Center (NCC), covers over 1400 hospitals across 31 provinces and over 10 million cancer patients in

Statistical and Epidemiological Analysis Plan (SEAP) for Observational and Non-Interventional Studies (ONIS)


China. This multicenter hospital-based database consists of data of 1509 variables from 7 aspects including drug, patient basic information, inpatient, outpatient, tests and examinations, treatment and follow up. NATDSS is linked with National Mortality Database from Chinese Center for Disease Control and Prevention Center (China CDC) to obtain patients' death information [R23-1183].

### 9. DATA MANAGEMENT AND SOFTWARE/TOOLS

#### 9.1 SOURCE DATA

Source data from the NATDSS are collected via an automatic web-based system, coded, deidentified and transmitted in a secure manner to maintain patient confidentiality compliant with national privacy standards. Source data will be desensitized by hiding the personal identifiable information or other sensitive information to create an Enterprise Master Patient Index (EMPI), which will allow individual level data to be linked when multiple sources are involved in the data integration process.

Authorization from NCC and Independent Ethics Committee (IEC) approval of leading site will be applied to ensure that the data are accessible and continuously active during study period.

#### 9.2 DATA CURATION

The data curation processes for this ONIS will be divided into the following parts.

- CRF generation: will design the first draft of variable list (CRF) and ensure that CRF is adequate for the collection of all relevant clinical data specified in the study protocol. CRF will be finalized after BI study team's review and confirmation.
- Data extraction: Scope of source data will be identified and extracted based on CRF and extraction plan. Data engineer from will verify critical parameters, including whether the data modules are complete, whether information for data encoding and decoding is clear, whether the mark of the data association is correct, whether the amount and characteristics of patients meet the requirements of the protocol, etc.
- Source data quality control: The source data will be evaluated across several aspects, including whether the data extraction is complete, whether the data conforms to the basic logic of medical records, and whether the threshold conforms to the normal clinical range. Regarding the data of logical value, abnormal value, and missing value, an effective data processing scheme shall be put forward. For any modification in the input process, confirmation and signature from the data engineer, as well as the reasons for the modification are required, to ensure that a complete audit trail has remained.
- Data transformation to project dataset: After data extraction is completed, multi-source data will be further standardized based on this study's design. Rules and procedures of data transformation will be reviewed and verified by medical experts and data engineers. Clinical information related to the same variable written in different terms will be standardized, normalized, and processed with logic and reasoning in medicine. The data management team will conduct a logic check on the entire finalized dataset after the extraction, where key data errors that can potentially affect this study will be corrected

Statistical and Epidemiological Analysis Plan (SEAP) for Observational and Non-Interventional Studies (ONIS)


through appropriate procedures. Finally, the structured and standardized data will be examined by trained reviewers, and then reviewed and signed by data manager. After the data is transformed, a sample of subjects will be selected to compare with source data for double-check.

Locking of project datasets: The dataset will be locked after all data quality control
processes are met. Any update needed for the locked dataset must be approved by the data
manager and processed appropriately in accordance with the standard dataset unlocking
process.

For this study, BI will not have access to the original data. Data will be managed by Source code of data management and data analyses will be stored for at least 15 years at .

#### 9.3 SOFTWARE/TOOLS

All computations and generation of tables, listings and data for figures will be performed using Statistical Analysis System (SAS) version 9.4 or higher (SAS). Used language and packages will be reported in the final report.

#### 9.4 HANDLING OF MISSING VALUES

Missing data may be encountered due to the study's retrospective nature and unavailability of data in electronic medical records. The number and percentages of patients with missing data for each variable will be summarized and reported. Only partial missing dates will be imputed, and no replacement/imputation procedures will be used for defined variables.

Missing dates will be imputed as follows: If the day is missing and the month and year is complete, the day will be imputed as the 15th of the month. If day and month or year was missing, the date will not be imputed and will be reported as missing.

### 10. DATA ANALYSIS

The statistical analysis plan for the study is summarized below. This study will be descriptive in nature.

For continuous variables, they'll be descriptively summarized using the mean with the standard deviation (SD), the median with the interquartile range (IQR), and the maximum and minimum values, as appropriate.

For categorical variables, the numbers and proportions of patients in different categories of the variable will be reported. Missing values will be presented as counts and percentages but excluded from the denominator when calculating proportions, unless there are additional instructions specified.

For time-to-event variables, the number and percentage of patients with events and censoring

Statistical and Epidemiological Analysis Plan (SEAP) for Observational and Non-Interventional Studies (ONIS)


will be summarized. The median survival time and its 95% confidence interval (CI) will be calculated using the Kaplan–Meier (KM) method, and KM plots will be provided.

It is anticipated that sample sizes for variables may vary due to unknown or missing data in the database. The number of patients with missing data for each variable will be summarized and reported. With the exception of the imputation of partial missing date values, no other imputation of missing values will be undertaken; however, the impact of missing data on interpretation of findings will be acknowledged and discussed in the final study report.

For all analyses, data for patients will be censored when lost to follow-up (i.e., still alive as of their last visit prior to end of study period).

### 10.1 MAIN ANALYSIS

### 10.1.1 Analysis of primary objective

OS will be analyzed for Cohort 1. For OS calculation, the event time is the date of death recorded by the National Mortality Database from CDC. OS is defined as the time from initiation of 1L until the date of death due to any cause. Patients without death record during the study period will be censored at the last medical record during the study period.

OS will be estimated by the KM method to obtain median estimates with 95% CIs and IQRs for Cohort 1, calculated using the log-log transformation. OS rate at 6, 12, 18, and 24 months will be described according to the survival curves if reached.

OS may be assessed by LOT and type of treatment received in each LOT, pending feasibility. OS by LOT is defined as the time from initiation of each LOT until the date of death due to any cause.

### 10.1.2 Analysis of secondary objectives

Survival after initial diagnosis will be estimated by the KM method to obtain median estimates with 95% CIs and IORs for Cohort 1 and Cohort 2.

Treatment patterns for Cohort 1 and Cohort 2 will be described by the number of lines, count with percentage (%) of patients by treatment lines, type of therapy and therapy regimens in each line.

LOTs are defined by the temporal relationship and sequencing of treatment regimens by using the dates of initiation and discontinuation of chemotherapy, targeted therapy, and/or immunotherapy. For each patient, 1L treatment regimen is defined as the first systemic treatment of any chemotherapy, and/or targeted drugs given to a patient after advanced or metastatic DDLPS diagnosis. A treatment line is advanced to the next line when a patient initiates new combinations of drugs or has the evidence of progression of disease. The start date of each LOT is defined as the date of initiation of new regimen, and the end date of each LOT is defined as the date of last dose prescribed or recorded at/before discontinuation.

Statistical and Epidemiological Analysis Plan (SEAP) for Observational and Non-Interventional Studies (ONIS)


### 10.3 SAFETY ANALYSIS

Not applicable.

Statistical and Epidemiological Analysis Plan (SEAP) for Observational and Non-Interventional Studies (ONIS)


### 11. QUALITY CONTROL

The study will strictly follow key elements of the Guideline for Good Pharmacoepidemiology Practices (GPP) and other relevant standard operating procedures (SOPs). The study report will be reviewed, approved and archived per BI SOP. Quality control methods during the whole process of data management is described in section 9, and quality control methods for data analyses are summarized below.

One data analyst from will build measures (variables) for cohort inclusion and outcomes. Whenever possible, validated algorithms will be used for variables, to minimize misclassification and information bias. All measures created, cohorts developed, statistical analyses implemented, and tables output will undergo quality control review performed by at least one additional Analyst from Quality controls include checks for the validity and logical content of codes and checks for missing values and variables. In order to control for potential inconsistencies and errors, all variables will be tabulated. The distribution of each variable will be examined.

The ONIS Lead will verify that the data analyst has followed methodology specified in the protocol, as well as any relevant programming SOPs and good programming practices. Documentation of key programming decisions should be evident within the program. The investigator or ONIS Lead will verify that any assumptions made by the data analyst are consistent with expectations.

### 12. REFERENCES

R14-4775

#### 12.1 PUBLISHED REFERENCES

| Care. |
|---------------|
| 5, |
| Liu, |
| ng |
| ;e |
| C |
| L<br>ng<br>ge |

Quan H, Sundararajan V, Halfon P, et al. Coding algorithms for defining

#### 12.2 UNPUBLISHED REFERENCES

Not applicable.

Statistical and Epidemiological Analysis Plan (SEAP) for Observational and Non-Interventional Studies (ONIS)


### ANNEX 1. ADDITIONAL INFORMATION

None.

### ANNEX 2. MOCK TABLE AND FIGURE

The following figures and tables will be developed for analyses of primary, secondary and exploratory objectives and will be replicated for subgroup analyses and sensitivity analyses, pending feasibility.

Table 1. Patient baseline demographic characteristics for Cohort 1 and Cohort 2

| Demographic characteristics | Cohort 1 | Cohort 2 |
|-----------------------------------------------|----------|----------|
| Number of patients, N | | |
| Index year, N (%)<br>2013 | | |
| 2014 | | |
| 2015 | | |
| 2016 | | |
| 2017 | | |
| 2018 | | |
| 2019 | | |
| 2020 | | |
| 2021 | | |
| Age at initial diagnosis, years | | |
| $Mean \pm SD$ | | |
| Median (IQR) | | |
| Min, Max | | |
| Missing / Unknown | | |
| Age (categorized) at initial diagnosis, N (%) | | |
| <65 | | |
| ≥65 | | |
| Missing / Unknown | | |
| Age at index, years | | |
| $Mean \pm SD$ | | |
| Median (IQR) | | |
| Min, Max | | |

Statistical and Epidemiological Analysis Plan (SEAP) for Observational and Non-Interventional Studies (ONIS)


| Demographic characteristics | Cohort 1 | Cohort 2 |
|-----------------------------------|----------|----------|
| Missing / Unknown | | |
| Age (categorized) at index, N (%) | | |
| <65 | | |
| ≥65 | | |
| Missing / Unknown | | |
| Sex, N (%) | | |
| Female | | |
| Male | | |
| Missing / Unknown | | |
| Insurance type, N (%) | | |
| National medical insurance | | |
| Commercial insurance | | |
| Out of pocket | | |
| Others | | |
| Missing / Unknown | | |
| Region, N (%) | | |
| Eastern China | | |
| Central China | | |
| Western China | | |
| Northeast China | | |
| Missing / Unknown | | |

Abbreviations: N = number; SD = standard deviation; IQR = interquartile range; min = minimum; max = maximum

Notes: Eastern China includes Beijing, Tianjin, Hebei, Shanghai, Jiangsu, Zhejiang, Fujian, Shandong, Guangdong, and Hainan; central China includes Shanxi, Anhui, Jiangxi, Henan, Hubei, and Hunan; western China includes Inner Mongolia, Guangxi, Chongqing, Sichuan, Guizhou, Yunnan, Tibet, Shaanxi, Gansu, Qinghai, Ningxia, and Xinjiang; northeast China includes Liaoning, Jilin, and Heilongjiang.

Statistical and Epidemiological Analysis Plan (SEAP) for Observational and Non-Interventional Studies (ONIS)


### Table 2. Patient clinical characteristics for Cohort 1 and Cohort 2

| Clinical characteristics | Cohort 1 | Cohort 2 |
|---|---|---|
| Number of patients, N<br>Year of initial diagnosis, N (%) | | |
| Before 2013 | | |
| 2013 | | |
| 2014 | | |
| 2015 | | |
| 2016 | | |
| 2017 | | |
| 2018 | | |
| 2019 | | |
| 2020 | | |
| 2021 | | |
| Missing / Unknown | | |
| Disease stage at initial diagnosis, N (%) | | |
| 0 | | |
| I | | |
| II | | |
| III | | |
| IV | | |
| Missing / Unknown | | |
| Histology, N (%) | | |
| Dedifferentiated | | |
| Other | | |
| Missing / Unknown | | |
| ECOG performance status, N (%) | | |
| 0 | | |
| 1 | | |
| 2 | | |
| 3 | | |
| 4 | | |
| Missing / Unknown | | |

Statistical and Epidemiological Analysis Plan (SEAP) for Observational and Non-Interventional Studies (ONIS)


| Clinical characteristics | Cohort 1 | Cohort 2 |
|---------------------------------|----------|----------|
| Primary tumor site, N (%) | | |
| Head or neck | | |
| Retroperitoneum or abdomen | | |
| Extremity | | |
| Pelvis | | |
| Thorax or trunk | | |
| Other | | |
| Missing / Unknown | | |
| Presence of metastases, N (%) | | |
| Yes | | |
| No | | |
| Missing / Unknown | | |
| Metastatic site, N (%) | | |
| Adrenal | | |
| Bone | | |
| Brain | | |
| Distant lymph node metastases | | |
| Liver | | |
| Lung | | |
| Other | | |
| Missing / Unknown | | |
| Number of surgeries prior to 1L | | |
| $Mean \pm SD$ | | |
| Median (IQR) | | |
| Min, Max | | |
| Missing / Unknown | | |
| Charlson comorbidity index | | |
| $Mean \pm SD$ | | |
| Median (IQR) | | |
| Min, Max | | |
| Missing / Unknown | | |
| History of smoking, N (%) | | |

Statistical and Epidemiological Analysis Plan (SEAP) for Observational and Non-Interventional Studies (ONIS)


| Clinical characteristics | Cohort 1 | Cohort 2 |
|--------------------------|----------|----------|
| Never smoker | | |
| Former smoker | | |
| Current smoker | | |
| Missing / Unknown | | |
| $BMI, kg/m^2$ | | |
| $Mean \pm SD$ | | |
| Median (IQR) | | |
| Min, Max | | |
| Missing / Unknown | | |

Abbreviations: N = number; SD = standard deviation; IQR = interquartile range; min = minimum; max = maximum; BMI = body mass index (defined as [weight in kilograms] / [height in meters]<sup>2</sup>); ECOG = Eastern Cooperative Oncology Group; 1L = first line.

Statistical and Epidemiological Analysis Plan (SEAP) for Observational and Non-Interventional Studies (ONIS)


#### Table 3. Overall survival from index for Cohort 1

At 18 months, [95% CI]

At 24 months, [95% CI]

| | Cohort 1 |
|---|---|
| | N= |
| Overall survival from Index, months | |
| KM Median, [95% CI] | |
| IQR | |
| Survival rate at different time point, (100/1000 person years)<br>At 6 months, [95% CI] | |
| At 12 months, [95% CI] | |

Abbreviations: KM= Kaplan–Meier; CI = confidence interval; IQR = interquartile range.

Statistical and Epidemiological Analysis Plan (SEAP) for Observational and Non-Interventional Studies (ONIS)


Table 4. Survival from initial diagnosis for Cohort 1 and Cohort 2

| | Cohort 1, | Cohort 2, |
|---|---|---|
| | <b>N</b> = | N= |
| Survival from initial diagnosis, months | | |
| KM Median, [95% CI] | | |
| IQR | | |
| Survival rate at different time point, (100/1000 person years)<br>At 6 months, [95% CI] | | |
| At 12 months, [95% CI] | | |
| At 18 months, [95% CI] | | |
| At 24 months, [95% CI] | | |

Abbreviations: KM= Kaplan–Meier; CI = confidence interval; IQR = interquartile range.

Statistical and Epidemiological Analysis Plan (SEAP) for Observational and Non-Interventional Studies (ONIS)


| Table 5. | Number | of total | lines of | f systemic | treatment |
|----------|--------|----------|----------|------------|-----------|

| | Cohort 1, | Cohort 2, |
|-----------------------------------------------|-----------|-----------|
| | N= | N= |
| Total lines of systemic treatment | | |
| $Mean \pm SD$ | | |
| Median (IQR) | | |
| Min, Max | | |
| Missing / Unknown | | |
| Total lines of treatment (categorized), N (%) | | |
| 1 | | |
| 2 | | |
| 3 | | |
| 4 | | |
| ≥5 | | |
| Missing / Unknown | | |

Abbreviations: N = number; SD = standard deviation; IQR = interquartile range; min = minimum; max = maximum.

Statistical and Epidemiological Analysis Plan (SEAP) for Observational and Non-Interventional Studies (ONIS) 

Table 6. Treatment types for Cohort 1 and Cohort 2 by line of therapy

| V 1 | Cohort 1, | | | | Cohort 2, | | |
|-----|-----------|----|----|---|------------|----|----|
| | N= | | | | <b>N</b> = | | |
| | 1L | 2L | 3L | _ | 1L | 2L | 3L |

Treated, N (%)

Yes

No

### Regimens, N (%)

Doxorubicin

Epirubicin

Liposomal doxorubicin

AD (doxorubicin, dacarbazine)

AIM (doxorubicin, ifosfamide, mesna)

Ifosfamide, epirubicin, mesna

Larotrectinib (NTRK fusion pos sarcomas only)

Entrectinib (NTRK fusion pos sarcomas only)

Pazopanib

Eribulin

Trabectedin

AD LMS only (doxorubicin, dacarbazine)

Gemcitabine and docetaxel

Gemcitabine

Gemcitabine and vinorelbine

Gemcitabine and dacarbazine

Dacarbazine

Ifosfamide

Temozolomide

Vinorelbine

Regorafenib

MAID (mesna, doxorubicin, ifosfamide, dacarbazine)

Statistical and Epidemiological Analysis Plan (SEAP) for Observational and Non-Interventional Studies (ONIS)


| | Cohort 1, | | | Cohort 2, | |
|---|-----------|------------|----|-----------|----|
| | | <b>N</b> = | | | N= |
| · | 1L 2L 3L | | 1L | 2L | 3L |

Pembrolizumab

durvalumab

Other

Concurrent steroid therapy, N (%)

Yes

No

Concurrent immunosuppressant therapy, N (%)

Yes

No

Concurrent hormone replacement therapy, N (%)

Yes

No

Abbreviations: 1L = first line; 2L = second line; 3L = third line.

Notes: Specific treatments and categories are ordered from highest to lowest frequency and may change upon examination of the data.

Statistical and Epidemiological Analysis Plan (SEAP) for Observational and Non-Interventional Studies (ONIS)


| Table 7. Time to next treatment | by l | line of | f treatment f | for | Cohort 1 | and | Cohort 2 |
|---|---|---|---|---|---|---|---|
|---|---|---|---|---|---|---|---|

| | Cohort 1, | Cohort 2, |
|---|---|---|
| | <b>N</b> = | N= |
| Treated, N (%) | | |
| Yes | | |
| No | | |
| Time from diagnosis to 1L treatment, months<br>Median, [95% CI] | | |
| IQR | | |
| Fime from 1L treatment to 2L treatment, months<br>Median, [95% CI] | | |
| IQR | | |
| Time from 2L treatment to 3L treatment, months<br>Median, [95% CI] | | |
| IQR | | |

Abbreviations: CI = confidence interval; IQR = interquartile range; 1L = first line; 2L = second line; 3L = third

Statistical and Epidemiological Analysis Plan (SEAP) for Observational and Non-Interventional Studies (ONIS)


| Table 8. Duration | of treatment by | line for | Cohort 1 | and Cohort 2 |
|-------------------|-----------------|----------|----------|--------------|

| | Cohort 1, | Cohort 2,<br>N= |
|----------------------------------|------------|-----------------|
| | <b>N</b> = | |
| Treated, N (%) | | |
| Yes | | |
| No | | |
| Duration of 1L treatment, months | | |
| Median, [95% CI] | | |
| IQR | | |
| Duration of 2L treatment, months | | |
| Median, [95% CI] | | |
| IQR | | |
| Duration of 3L treatment, months | | |
| Median, [95% CI] | | |
| IQR | | |

Abbreviations: CI = confidence interval; IQR = interquartile range; 1L = first line; 2L = second line; 3L = third line.

Statistical and Epidemiological Analysis Plan (SEAP) for Observational and Non-Interventional Studies (ONIS)


Table 9. Healthcare resource utilization for Cohort 1 and Cohort 2

| | Cohort 1, | Cohort 2, |
|---|---|---|
| | N= | N= |
| Inpatient admissions | | |
| $Mean \pm SD$ | | |
| Median (IQR) | | |
| Min, Max | | |
| Missing / Unknown | | |
| Total days of hospital stay for inpatien $\operatorname{Mean} \pm \operatorname{SD}$ | nt admission, days | |
| Median (IQR) | | |
| Min, Max | | |
| Missing / Unknown | | |
| Average days of hospital stay for each Mean $\pm$ SD | inpatient admission, days | |
| Median (IQR) | | |
| Min, Max | | |
| Missing / Unknown | | |
| Outpatient visits | | |
| $Mean \pm SD$ | | |
| Median (IQR) | | |
| Min, Max | | |
| Missing / Unknown | | |
| Emergency room visits | | |
| $Mean \pm SD$ | | |
| Median (IQR) | | |
| Min, Max | | |
| Missing / Unknown | | |

Abbreviations: SD = standard deviation; IQR = interquartile range; min = minimum; max = maximum

Table 10. Direct medical cost for Cohort 1 and Cohort 2

| | Cohort 1, | Cohort 2, |
|---|---|---|
| | <b>N</b> = | N= |
| Total cost of hospitalization, CNY $Mean \pm SD$ | | |
| Median (IQR) | | |
| Min, Max | | |
| Missing / Unknown | | |
| Average cost per hospitalization, CNY $Mean \pm SD$ | | |
| Median (IQR) | | |
| Min, Max | | |
| Missing / Unknown | | |
| Total cost of outpatient visit, CNY $Mean \pm SD$ | | |
| Median (IQR) | | |
| Min, Max | | |
| Missing / Unknown | | |
| Average cost per outpatient visit, CNY $Mean \pm SD$ | | |
| Median (IQR) | | |
| Min, Max | | |
| Missing / Unknown | | |
| Total cost of Emergency Room visit, CNY $Mean \pm SD$ | | |
| Median (IQR) | | |
| Min, Max | | |
| Missing / Unknown | | |
| Average cost per Emergency Room visit, CNY $\label{eq:mean} \mathbf{Mean} \pm \mathbf{SD}$ | | |
| Median (IQR) | | |
| Min, Max | | |
| Missing / Unknown | | |

Abbreviations: SD = standard deviation; IQR = interquartile range; min = minimum; max = maximum; CNY = Chinese Yuan

Statistical and Epidemiological Analysis Plan (SEAP) for Observational and Non-Interventional Studies (ONIS)

Figure 1. Kaplan-Meier curve of Overall survival for Cohort 1, from index



Figure 2. Kaplan-Meier curve of survival after initial diagnosis for Cohort 1 and Cohort 2, from initial diagnosis



Statistical and Epidemiological Analysis Plan (SEAP) for Observational and Non-Interventional Studies (ONIS)

Figure 3. Kaplan-Meier curve of time to next treatment for Cohort 1 and Cohort 2, from 1L initiation



Statistical and Epidemiological Analysis Plan (SEAP) for Observational and Non-Interventional Studies (ONIS)


Figure 4. Kaplan-Meier curve of duration of treatment for Cohort 1 and Cohort 2, from 1L initiation

